CLINICAL TRIAL: NCT02387697
Title: Treatment of Severe Secondary TRIcuspid Regurgitation in Patients With Advance Heart Failure With CAval Vein Implantation of the Edwards Sapien XT VALve
Brief Title: Treatment of Severe Secondary TRIcuspid Regurgitation in Patients With Advance Heart Failure With CAval Vein Implantation of the Edwards Sapien XT VALve (TRICAVAL)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Karl Stangl, Prof. Dr. med Karl Stangl, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRICAVAL
Record Dates: First submitted 2015-02-27; First posted 2015-03-13 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Severe Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Transfemoral implantation of an Edwards Sapien XT Valve into the vena cava inferior (VCI). For better stability and for downsizing of the VCI diameter the valve will be implanted after preparation of a landing zone. This includes implantation of one or two self expandable stents into the VCI prior to the final deployment of the valve.
  Interventions: Device: Edwards Sapien XT Valve
- Group B (No Intervention): Control group (no surgery) with optimal medical treatment.

INTERVENTIONS:
Device: Edwards Sapien XT Valve — The device will be implanted in the present study to prevent abdominal venous congestion and to improve the function of the tricuspid valve which is located in the low pressure system in the right heart.
  Arms: Group A

SUMMARY:
The purpose of this study is to assess the efficacy and safety of implanting an Edwards Sapien XT Valve into the vena cava inferior (VCI; between right atrium and the hepatic vein) on clinical variables, exercise tolerance and well being in patients with severe tricuspid regurgitation and signs of right heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic tricuspid regurgitation with a significant regurgitation jet into the caval and hepatic veins
* Optimal medical treatment
* High surgical risk with STS Score ≥ 10 or logistic EuroSCORE I ≥ 15 or any contraindication for conventional valve replacement/repair
* NYHA class of at least II
* Written informed consent

Exclusion Criteria:

* VCI diameter > 32 mm
* Severe left ventricular dysfunction with LVEF < 30%
* Severe mitral insufficiency
* Estimated life expectancy < 12months (360 days) due to carcinoma, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease
* Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment
* Evidence of stroke / TIA during the last 180 days
* Leukopenia (WBC < 3000 cell/mL), anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cells/mL), or any known blood clotting disorder
* Evidence of an intracardiac mass, thrombus or vegetation
* Active upper GI bleeding within 1 month (30 days) prior to procedure
* Patients with an acute emergency
* Contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure
* Allergy against the use of implanted stent / prosthesis
* Patient undergoing regular dialysis or a serum creatinine above 3.0 mg/dl
* Patients unsuitable for implantation because of thrombosis of the lower venous system or vena cava filter
* Active bacterial endocarditis within 6 months (180 days) of procedure.
* Women of childbearing potential without highly effective contraception (PEARL-Index < 1%)
* Inability to comply with all of the study procedures and follow-up visits
* Subjects who are legally detained in an official institute (according to § 20 MPG)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximum relative VO2 uptake | at 3 month
  we consider the difference of means in maximum relative VO2 uptake at 3 months compared to control group.

SECONDARY OUTCOMES:
NYHA class | day 30 and month 3
ejection fraction (EF) | day 30 and month 3
right ventricular (RV) diameter | day 30 and month 3
right atrial (RA) diameter | day 30 and month 3
hepatic vein diameter | day 30 and month 3
N-terminal pro Brain Natriuretic Peptide (NT-proBNP) | day 30 and month 3
tricuspid regurgitation jet velocity time integral (as assessed by Doppler echocardiography) | day 30 and month 3
aerobic threshold (assessed by spiroergometry) | day 30 and month 3
ventilation efficiency (as assessed by the VE / VCO2 slope in spiroergometry) | day 30 and month 3
Unscheduled rehospitalization | day 30 and month 3
Dyspnoea VAS | day 30 and month 3
Minnesota Living with Heart Failure Questionnaire | day 30 and month 3
6-minutes walk test | day 30 and month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Charite Universitaetsmedizin, Medizinische Klinik für Kardiologie und Angiologie, Berlin, Germany

REFERENCES:
- [Derived] Mattig I, Hewing B, Knebel F, Meisel C, Ludwig A, Konietschke F, Stangl V, Stangl K, Laule M, Dreger H. Effect of inferior caval valve implantation on circulating immune cells and inflammatory mediators in severe tricuspid regurgitation. BMC Cardiovasc Disord. 2024 Jul 18;24(1):373. doi: 10.1186/s12872-024-04044-1. PMID 39026154